CLINICAL TRIAL: NCT04902092
Title: Brain Exercise and Addiction Trial: Efficacy of a 12-week Aerobic Exercise Regime for Restoring 'Brain Health' in Cannabis Users
Brief Title: Brain Exercise and Addiction Trial
Acronym: BEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: Turning Point (Other)
Responsible Party: Principal Investigator, Rebecca Segrave, Senior Research Fellow, Monash University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12563
Record Dates: First submitted 2021-05-13; First posted 2021-05-26 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Cannabis Use Disorder, Moderate; Cannabis Use Disorder, Severe
MeSH Terms: conditions — Lymphoma, Follicular | interventions — High-Intensity Interval Training; Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Physical Training (Active Comparator): 12-week, 36 session, cardiorespiratory-focussed physical exercise program delivered by an accredited exercise physiologist
  Interventions: Behavioral: High Intensity Interval Training
- Low Intensity Physical Training (Active Comparator): 12- week, 36 session, strength-focussed physical exercise program delivered by an accredited exercise physiologist
  Interventions: Behavioral: Strength and Resistance Training

INTERVENTIONS:
Behavioral: High Intensity Interval Training — Exercise sessions will commence with an initial 3-week accustomization period whereby training load will increase incrementally from 2 x 45min sessions with effort peaking at 60% VO2 max (week 1) increasing to 3 x 45minute with effort peaking at 80% VO2max (week 3). Participants will transition to the full HIIT protocol for the remaining weeks. The HIIT component will comprise a work-rest ratio of ≥1:1minutes, with alternating exertion epochs at >80% VO2max and <60% VO2max. As VO2max is likely to increase as fitness improves toward the end of the 3-month program, adjustments to HIIT will be made by the exercise physiologist based on real-time heart rate monitoring, ensuring greater accuracy in participants achieving their heart rate targets.
  Arms: High Intensity Physical Training
Behavioral: Strength and Resistance Training — Exercise sessions will comprise a combination of strength, coordination and mobility exercises. The strength component will consist of 2-3 sets of resistance exercises at ≤70% of a predicted 1 repetition maximum, targeting all body segments. Heart rate tracking will occur to ensure participants do not exceed 70% v02 (or exceed Lactate Threshold).
  Arms: Low Intensity Physical Training

SUMMARY:
Heavy cannabis use is associated with substantive learning and memory impairments and elevated risk of psychopathology. It has been repeatedly demonstrated that the hippocampus, centrally implicated in these processes, is particularly vulnerable to the deleterious effects of prolonged exposure to cannabis. This deterioration of hippocampal structure, function, and biochemistry can be reversed, but this requires two or more years of abstinence from cannabis. However, most heavy cannabis users find it extremely difficult to maintain abstinence over extended periods and current treatments for cannabis use disorders are inadequate. There is a pressing clinical need for an intervention that rapidly accelerates hippocampal recovery, ameliorates the associated cognitive impairments and mental health symptoms, and leads to improved treatment outcomes. One promising candidate is physical exercise. In addition to the well-known physical health benefits, regular exercise also has a potent positive effect on brain health. The current study will investitive the capacity of two different neuroscientifically-informed 12-week exercise programs can restore brain health for heavy long term cannabis users.

DETAILED DESCRIPTION:
Heavy cannabis use is associated with substantive learning and memory impairments and elevated risk of psychopathology. It has been repeatedly demonstrated that the hippocampus, centrally implicated in these processes, is particularly vulnerable to the deleterious effects of prolonged exposure to cannabis. This deterioration of hippocampal structure, function, and biochemistry can be reversed, but this requires two or more years of abstinence from cannabis. However, most heavy cannabis users find it extremely difficult to maintain abstinence over extended periods and current treatments for cannabis use disorders are inadequate. There is a pressing clinical need for an intervention that rapidly accelerates hippocampal recovery, ameliorates the associated cognitive impairments and mental health symptoms, and leads to improved treatment outcomes. One promising candidate is physical exercise. In addition to the well-known physical health benefits, regular exercise also has a potent positive effect on brain health and can increase the size of the hippocampus. It's not yet known how much or what kind of exercise produces the best results. This study has been designed to compare the effects of two different exercise programs.

1. 12 weeks of regular HIIT exercise
2. 12 weeks of regular strength training

The research team are investigating whether the programs have a positive impact on brain health and, if they do, whether one is more effective than the other. The research team will also measure whether engaging in either program leads to a reduction in cannabis consumption, and improvements in thinking skills, mental health, and general wellbeing.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20-55 years
2. Voluntary and able to provide informed consent
3. Fluent in English
4. Current moderate - severe cannabis use disorder
5. Major history of cannabis use (i.e. ≥3 days per week on average for ≥4 of the past 6 years)
6. Capacity to tolerate physical exercise according to 'Fitness to Exercise'

Exclusion Criteria:

1. Have a history of cardiovascular disease, high blood pressure, musculoskeletal injury or other condition that would preclude safe engagement in VO2 max fitness testing and/or regular physical exercise
2. Severe claustrophobia, non-MR compatible metallic implant, or other contraindication to MRI scanning
3. Lifetime history of significant neurological illness, or moderate - severe brain injury,
4. Current major unstable medical illness or chronic pain condition
5. Lifetime history of schizophrenia, schizoaffective disorder, OCD, PTSD, bipolar disorder
6. Current significant depression or anxiety that precludes ability to reliably engage in the exercise program
7. Current moderate - severe substance use disorder for substances other than cannabis (excluding nicotine)
8. Currently pregnant or lactating
9. Shift work employment schedule within the prior 6-months
10. Have engaged in ≥5 sessions of HITT or resistance training within the past 12-months
11. History of treatment with antipsychotic medications
12. Current participation in psychosocial treatment for substance use disorder
13. Other psychoactive medications or psychosocial treatments will be considered on a case-by-case basis. Where a current psychoactive medication is deemed acceptable, both dose and type must have been stable for a minimum of four weeks prior to baseline assessment, and remain stable throughout the 12-week exercise phase of the study.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Change in hippocampal integrity | Baseline (0 months), post (3 months)
  Composite score derived from three hippocampal health indices: volume (structural MRI), connectivity (DTI), neuronal health (MRS NAA) calculated as described in Yucel et al (2016), doi:10.1038/tp.2015.201.

SECONDARY OUTCOMES:
Change in cannabis use | Baseline (0 months), post (3 months), follow up (6 months)
  Time line follow back
Change in cannabis dependence | Baseline (0 months), post (3 months), follow up (6 months)
  Severity of Dependence Scale (SDS; range = 0-15 higher scores indicate higher dependence
Change in cannabis craving | Baseline (0 months), post (3 months), follow up (6 months)
  Penn Craving Scale (PCS; range = 0 - 30 higher scores indicate greater craving)
Change in depression symptoms | Baseline (0 months), post (3 months), follow up (6 months)
  Quick Inventory of Depressive Symptomology (QUIDS; range = 0 - 27 higher scores indicate greater depression symptom severity)
Change in anxiety symptoms | Baseline (0 months), post (3 months), follow up (6 months)
  StateTrait Anxiety Inventory (STAI; range = 20 to 80, higher scores indicate greater anxiety)
Change in resilience | Baseline (0 months), post (3 months), follow up (6 months)
  Connor David Resilience Scale (CDRS; range = 0-100 higher scores indicate higher resilience)
Change in coping skills | Baseline (0 months), post (3 months), follow up (6 months)
  Perceived Stress Scale (10 item; range = 0 - 40 higher scores indicate greater stress)
Change in sleep quality | Baseline (0 months), post (3 months), follow up (6 months)
  Pittsburgh Sleep Quality Index (PSQI; range = 0 to 21 higher scores indicate worse sleep quality)
Change in mental wellbeing | Baseline (0 months), post (3 months), follow up (6 months)
  Warwick Edinburgh Mental Wellbeing Scale (WEMWBS; range = 14-70 higher scores indicate increased mental well being)
Change in quality of life | Baseline (0 months), post (3 months), follow up (6 months)
  Quality of Life and Satisfaction Questionnaire - Short Form (QOL-SF; range = 70 higher scores indicate greater life satisfaction and enjoyment)
Change in memory | Baseline (0 months), post (3 months), follow up (6 months)
  Rey Auditory Verbal Learning Test (RAVLT)
Change in associative memory | Baseline (0 months), post (3 months), follow up (6 months)
  Paired Associates Learning Task (PAL)
Change in visual memory | Baseline (0 months), post (3 months)
  Figural Memory Tasks
Change in cardiorespiratory fitness | Baseline (0 months), post (3 months)
  VO2 max

CONTACTS AND LOCATIONS:
Overall Officials: Murat Yucel, Principal Investigator — Monash University
Locations (1):
- Monash University, BrainPark, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Richardson KE, Suo C, Albertella L, Maleki S, Coxon J, Hendrikse J, Hughes S, Pitt J, Kayayan E, Brown C, Nguyen L, Solowij N, Lubman DI, Segrave R, Yucel M. High-Intensity Exercise and Hippocampal Integrity in Adults With Cannabis Use Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2025 Dec 1;82(12):1240-1245. doi: 10.1001/jamapsychiatry.2025.2319. PMID 40928796